CLINICAL TRIAL: NCT00374036
Title: Strategy Phase III Intergroup Study for Chemotherapy of the Metastatic or Locally Advanced Cancers of the Stomach
Brief Title: Metastatic Gastric Cancer FFCD 03-07
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Federation Francophone de Cancerologie Digestive (Other); Roche Pharma AG (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0305603
Record Dates: First submitted 2006-09-06; First posted 2006-09-08 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Stomach Cancer; Neoplasm Metastasis
Keywords: chemotherapy; stomach cancer metastatic; Capecitabine; Irinotecan
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis | interventions — IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): ECC
  Interventions: Drug: ECC
- 2 (Experimental): FOLFIRI
  Interventions: Drug: FOLFIRI

INTERVENTIONS:
Drug: ECC — capecitabine
  Arms: 1
Drug: FOLFIRI — Irinotecan
  Arms: 2

SUMMARY:
The purpose of this study is to compare the effectiveness of 2 different sequences of polychemotherapy among carrying patients of a adenocarcinoma of the stomach or cardia locally advanced or metastatic.

DETAILED DESCRIPTION:
To compare the effectiveness of two different sequences of polychemotherapy among carrying patients of a adenocarcinoma of the stomach or cardia locally advanced or metastatic.

ELIGIBILITY:
Inclusion Criteria:

* age = 18 years old
* patients carrying a adenocarcinoma of the stomach or cardia histologically proven
* locally advanced tumour which may not be treated surgically or metastatic tumour
* the patients having a stenosante tumour responsible for a disphagy had to have a tumoral ablation or a prosthesis or a probe of food,
* measurable lesions according to criteria RECIST (specify measurement by spiral scanner of largest diameter of with less the one lesion of size higher than 1 cm) or appraisable but nonmeasurable (lesions < 1 cm, ascite, pleural effusion...)
* general state WHO < 2
* absence of insufficiency cardiac or coronary symptomatic
* absence of previous chemotherapy other that auxiliary stopped since more than 6 months
* filled questionnaires QLQ C30 and STO-22
* PNN = 1500/mm3, haemoglobin ≥ 10g/dl, plates= 100 000/mm3
* creatinin ≤ 110 micromol/l
* bilirubin ≤ 35 micromol/l

Exclusion Criteria:

* disphagy or intestinal obstruction incompatible with a treatment per os or by a probe of food
* pregnant or nursing woman
* previous of cardiac toxicity to the 5FU or to the anthracyclines
* radiotherapy less than 3 weeks before inclusion, whatever the site
* other evolutionary cancer threatening the short-term life
* metastasis cerebral or méningée known (without obligation to seek it)
* impossibility of regular follow-up for psychological, social, family or geographical reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2005-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Time until therapeutic failure : to make pass TET from 15 weeks with ECC in first line to 20 weeks with FOLFIRI in first line | 20 weeks

SECONDARY OUTCOMES:
Time of total survival and survival without progression | 3 years
The percentage of objective answers in first and second line | 1 year
Percentage of treated patients in second line | 3 years
Control time of the disease | 3 years
The tolerance, the quality of life, duration of hospitalization | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Rosine GUIMBAUD, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France

REFERENCES:
- [Derived] Guimbaud R, Louvet C, Ries P, Ychou M, Maillard E, Andre T, Gornet JM, Aparicio T, Nguyen S, Azzedine A, Etienne PL, Boucher E, Rebischung C, Hammel P, Rougier P, Bedenne L, Bouche O. Prospective, randomized, multicenter, phase III study of fluorouracil, leucovorin, and irinotecan versus epirubicin, cisplatin, and capecitabine in advanced gastric adenocarcinoma: a French intergroup (Federation Francophone de Cancerologie Digestive, Federation Nationale des Centres de Lutte Contre le Cancer, and Groupe Cooperateur Multidisciplinaire en Oncologie) study. J Clin Oncol. 2014 Nov 1;32(31):3520-6. doi: 10.1200/JCO.2013.54.1011. Epub 2014 Oct 6. PMID 25287828